CLINICAL TRIAL: NCT02587117
Title: Comparative Study of the Efficacy of Lycopene Versus Prednisolone in the Management of Oral Lichen Planus: A Randomized, Double Blind Clinical Trial
Brief Title: A Clinical Trial to Study the Effects of Two Drugs, Lycopene and Prednisolone in Patients With Oral Lichen Planus
Acronym: OLP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Ramayan Prasad Kushwaha, assistant professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 636/069/070
Record Dates: First submitted 2015-10-20; First posted 2015-10-27 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Oral Lichen Planus
Keywords: Antioxidant; Lycopene; Prednisolone
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Lycopene; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lycopene group (Experimental): Lycopene- 4 mg capsule by mouth single dose per day for 2 months
  Interventions: Drug: lycopene
- Prednisolone group (Active Comparator): Prednisolone- 40 mg capsule by mouth single dose per day for 2 months
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: lycopene — Each capsule contain 2 mg lycopene. Each patient was received two capsules of lycopene (total dose was 4 mg) single dose in morning for 2 months. Follow-up was done at base line, 2nd, 4th, 6th and 8th weeks of the therapy.
  Other Names: lycored
  Arms: lycopene group
Drug: Prednisolone — Each capsule contain 20 mg prednisolone. Each patient was received two capsules of prednisolone (total dose was 40 mg) single dose in morning for 2 months. Follow-up was done at base line, 2nd, 4th, 6th and 8th weeks of the therapy.
  Other Names: wysolone
  Arms: Prednisolone group

SUMMARY:
Oral lichen planus (OLP) is a common sub-acute, chronic inflammatory mucocutaneous disease.This study was evaluated the comparative efficacy of lycopene and prednisolone for the treatment of oral lichen planus. Half of participants (total number of participants was twenty eight) were received lycopene and the other half were received prednisolone.

DETAILED DESCRIPTION:
Prednisolone and lycopene were produced remission of lesions in oral lichen planus patients, but they do so by different mechanisms.

The main cause of oral lichen planus is still unknown. Some authors advocate the disease appears to be a result of T-cell-mediated autoimmune responses in oral epithelial tissues. But, recent study suggests that increased reactive oxygen species (ROS) and lipid peroxidation together with an imbalance in the antioxidant defense system may play a part in the generation of disease.

Lycopene exerts its antioxidant activity by physical and chemical quenching of free radicals and decreases free radicals-initiated oxidative reactions, particularly lipid peroxidation and DNA oxidative damage, thereby preventing tissue damage.

Prednisone have both anti-inflammatory and immunosuppressant effects.It suppresses the inflammatory response by limiting the recruitment of inflammatory cells and inhibiting synthesis of pro-inflammatory products such as prostaglandins (PGs), leukotrienes (LTs) and platelet activating factors (PAF) by indirectly inhibiting phospholipase A2 and negative regulating cyclooxygenase (COX-2).

ELIGIBILITY:
Inclusion Criteria:

* Subject had symptomatic i.e. burning sensation and/or pain secondary to oral lichen planus.
* Subject had clinically & histo-pathologically diagnosed as oral lichen planus.
* Subject had not on any treatment for the same or treatment likely to modify their oral lichen planus (e.g. systemic steroids, antifungals, immunosuppressant's, anti-oxidant).

Exclusion Criteria:

* Suffering from any systemic disease/s such as diabetes, hypertension, cardiovascular, respiratory system disease, renal dysfunction, liver disorders, malignancy, active peptic ulcer diseases, acute gastrointestinal diseases, anemia and glaucoma, etc.
* Suffering from serious or recurrent infection, immunodeficiency or HIV.
* Pregnant or breast feeding (including women who wish to be pregnant during the study period).
* Any other mucosal diseases or any other skin diseases which might be associated with oral lesions.
* On any drug therapy which might be causes lichen planus like lesions.
* Known allergy or contraindication to study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramayan Pr Kushwaha, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences (BPKIHS), Dharan, Nepal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only symptomatic oral lichen planus patients, who were fulfill inclusion and exclusion criteria, were selected and recruited from the outpatient department of Oral Medicine and Radiology, College of dental surgery, BPKIHS on the basis of randomization list. The first patients was recruited on 21/02/2013 and the last patients was on 28/01/2014.
Pre-assignment Details: Before enrollment, full explanation about the study was given and written informed consent was taken. A detailed clinical history, clinical examination,baseline investigations and punch biopsy were taken. Patient was on treatment with medication for the same lesions asked to stop the treatment and a washout period of 3 weeks was given.
Period: Overall Study
Arm/Group | Lycopene Group | Prednisolone Group
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lycopene Group | Prednisolone Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.69 (13.97) | 48.07 (12.27) | 45.11 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 7 | 3 | 10
Piboonniyom REU (Reticular, Erythematous and Ulceration) severity score [Mean (Standard Deviation); unit: Scores on a scale] — Reticular:score 0=no white striations; score1= white striations. Erythematous:score 0=no lesion; score1= lesion <1 cm2; score2: lesion 1-3 cm2; score3= lesion >3 cm2. Ulceration:score 0=no lesion; score1= lesion <1 cm2; score2= lesion 1-3 cm2; score3= lesion >3 cm2. Total weighted score was sum total scores of each lesion & multiplication with weighted score 1.5 & 2.0 in total erythematous & total ulceration scores=ΣR+ΣE×1.5+ΣU×2.0. Total score was dependent on the number of lesions of each participant. Higher values of total score represent worse outcome & zero value represent no lesion.
  Scores on a scale | 8.23 (5.85) | 8.34 (7.83) | 8.28 (6.86)
Baseline NRS (numerical rating scale) burning sensation score [Mean (Standard Deviation); unit: Scores on a scale] — Each patient was provided standard self-response Numerical Rating Scale (NRS) of 0 (no oral discomfort) to 10 (worst imaginable oral discomfort) to respond the intensity of burning sensation or pain or discomfort during each visit. the mean of NRS burning sensation score was calculated and considered as baseline NRS burning sensation score.
  Scores on a scale | 3.69 (1.75) | 3.60 (2.03) | 3.64 (1.87)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Lesions(Degree of Reticular, Erythematous and Ulceration) by Using Piboonniyom REU Severity Score
Description: Reticular: score 0= no white striations; score 1= white striations. Erythematous: score 0= no lesion; score 1= lesion <1 cm2; score 2: lesion 1-3 cm2; score 3= lesion >3 cm2. Ulceration: score 0= no lesion; score 1= lesion <1 cm2; score 2= lesion 1-3 cm2; score 3= lesion >3 cm2. Total weighted score was derived by sum total scores of each lesion and multiplication with weighted score 1.5 & 2.0 in total erythematous and total ulceration scores as ΣR + ΣE × 1.5 + ΣU × 2.0.Total weighted score was dependent on the number of lesions of each participant which was not the same across participants. Higher value of the total score represent worse outcome & zero value represent no lesion.
Time Frame: 8 weeks minus baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lycopene Group | Prednisolone Group
Number analyzed (Participants) | 13 | 15
Scores on a scale | 2.15 (1.68) | 0.73 (1.58)
Statistical Analysis 1: Comparison: Lycopene Group vs Prednisolone Group; Test type: Superiority or Other; p = 0.004, Mann Whitney test

2. Secondary Outcome: Burning Sensation or Pain by Using NRS (Numerical Rating Scale)
Description: Standard self-response Numerical Rating Scale (NRS) of 0 (no oral discomfort) to 10 (worst imaginable oral discomfort) to represent the intensity of burning sensation or pain or discomfort. The mean of NRS burning sensation score was calculated after eight weeks of treatment and considered as 8th week NRS burning sensation score.
Time Frame: 8 weeks minus baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lycopene Group | Prednisolone Group
Number analyzed (Participants) | 13 | 15
Scores on a scale | 0.23 (0.44) | 0.07 (0.26)
Statistical Analysis 1: Comparison: Lycopene Group vs Prednisolone Group; Test type: Superiority or Other; p = 0.224, Mann Whitney test

ADVERSE EVENTS:
Time Frame: Daily monitoring throughout 8 weeks of treatment
Arm/Group | Lycopene Group | Prednisolone Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 10/13 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lycopene Group (N=13) | Prednisolone Group (N=15)
Puffiness of face (General disorders) | 0 (0) | 13 (13)
Headache (Nervous system disorders) | 1 (1) | 10 (10)
Dizziness (Nervous system disorders) | 1 (1) | 8 (8)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 6 (6)
Blurred vision (Eye disorders) | 0 (0) | 4 (4)
Flatulency (Gastrointestinal disorders) | 9 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to limitation of time, there were small numbers of subjects enrollment; not possible to follow-up the cases after the treatments were over and to determine the relapse rate of the patients; performed at a single medical center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes